CLINICAL TRIAL: NCT05633446
Title: A Phase I-II, Blinded, Randomized, Placebo-controlled Study of a T Cell Priming Next-generation Vaccine Against Coronavirus Disease in Healthy Adults
Brief Title: Next Generation T-cell Vaccine Against Coronavirus Disease (COVID-19)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gylden Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: naNO-COVID 2
Record Dates: First submitted 2022-11-30; First posted 2022-12-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Coronavirus; SARS-CoV-2 Infection; COVID-19
Keywords: Coronavirus; SARS-CoV-2; COVID-19; T-cell priming; COVID vaccine; Nanoparticle; T cell; Cellular immunity; T-cell vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: * This trial is double-blinded (blinded to investigators and participants)
  * Blinding will be maintained for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PepGNP-COVID19 (One vaccination) (Experimental): One vaccination of PepGNP-COVID19 vaccine candidate administered on Day 0 (50 µl per dose)
  Interventions: Biological: PepGNP-COVID19 (One vaccination)
- Placebo (One vaccination) (Placebo Comparator): One vaccination of WFI administered on Day 0 (50 µl per dose)
  Interventions: Other: Water for injection (One vaccination)
- PepGNP-COVID19 (Two vaccinations) (Experimental): Two vaccinations of PepGNP-COVID19 vaccine candidate administered on Day 0 and Day 21 (50 µl per dose)
  Interventions: Biological: PepGNP-COVID19 (Two vaccinations)
- Placebo (Two vaccinations) (Placebo Comparator): Two vaccinations of WFI administered with on Day 0 & Day 21 (50 µl per dose)
  Interventions: Other: Water for injection (Two vaccinations)

INTERVENTIONS:
Biological: PepGNP-COVID19 (One vaccination) — One dose with 7.5 nmol total peptide/dose with 47.8ug gold base particle in 50 µl WFI
  Arms: PepGNP-COVID19 (One vaccination)
Other: Water for injection (One vaccination) — Water For Injection (WFI): (sodium chloride, a 0.9% solution for the preparation of dosage forms for injections) 50 µl per dose
  Other Names: WFI
  Arms: Placebo (One vaccination)
Biological: PepGNP-COVID19 (Two vaccinations) — Two vaccinations with 7.5 nmol total peptide/dose with 47.8ug gold base particle in 50 µl WFI
  Arms: PepGNP-COVID19 (Two vaccinations)
Other: Water for injection (Two vaccinations) — Water For Injection (WFI): (sodium chloride, a 0.9% solution for the preparation of dosage forms for injections) 50 µl per dose
  Other Names: WFI
  Arms: Placebo (Two vaccinations)

SUMMARY:
The study aims to investigate the safety and immunogenicity of one dose vs two doses of a T-cell priming next-generation vaccine against Coronavirus disease.

DETAILED DESCRIPTION:
The scale of the COVID-19 pandemic requires multiple vaccine candidates to ensure equitable and rapid access to protection by:

* Providing a range of vaccine choices tailored to variations in immunological profiles across demographics as well as suited to environments with various levels of resources (cold chain etc).
* Distributing and parallelizing manufacture, to speed up scale, avoid reagent stockouts and dilute monopolies

  * The ability for SARS -CoV-2 (Severe Acute Respiratory Syndrome Coronavirus-2) to mutate, requires multiple vaccine candidates to ensure robust and sustainable protection. Vaccines with a range of epitopes and immune targets provide immunological diversity and reduce vulnerability to mutant escape.
  * Nanotechnology fulfils the needs of a Universal Coronaviruses vaccine by being a rapidly scalable and modular platform
  * Humoral immunity may be transient and insufficient against emerging variants of SARS-CoV-2
  * Cellular immunity against SARS-CoV-2 is lasting and associated with recovery in COVID-19. A vaccine (prime or booster) inducing the right T cell response can be the solution against the need to develop new vaccines every time the virus mutates or a new variant persists.

This is a Phase I-II, double-blind, randomized, placebo-controlled study investigating the safety and immunogenicity of a T cell priming next-generation vaccine against Coronavirus disease in healthy adults.

The clinical study will enrol 110 participants (88 vaccine vera and 22 placebo, [split 50:50 between two groups one receiving one vaccination and the other two vaccinations]).

Therefore, 110 eligible participants will be randomized in the following groups:

* Group 1 One Vaccination (Day 0) (n=55): 44 PepGNP-COVID19 (7.5 nmol peptide + 47.8ug GNP) + 11 placebo (WFI)
* Group 2 Two Vaccinations (Day 0 & Day 21) (n=55): 44 PepGNP-COVID19 (7.5 nmol peptide + 47.8ug GNP) + 11 placebo (WFI) Allocations of vaccine vera vs placebo for each group are single blinded."

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18 to 75 years on the day of inclusion
2. Participant signed informed consent
3. Residing in Philippines.
4. A participant can be included providing COVID-19 polymerase chain reaction (PCR) test is negative at screening.
5. A participant can be included providing, the participant haven't received any vaccination against COVID-19 in the past, or if the participant had already received any of the following licensed vaccines against COVID-19: Oxford/AstraZeneca; Pfizer/BioNTech; Moderna; or J&J/Janssen, with the participants last dose received at least 6 months prior the inclusion in this trial.

Exclusion Criteria:

1. Participant is pregnant, lactating, or of childbearing potential
2. Participation in the 6 months preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
3. Receipt of any vaccination against COVID-19 less than 6 months prior to participation in study.
4. Receipt of any vaccine in the three months preceding the first trial vaccination or planned receipt of any vaccine in the 6 months following last trial vaccination.
5. Positive SARS-CoV-2 test in the 4 weeks preceding the first trial vaccination
6. Receipt of immunoglobulins, blood, or blood-derived products in the past 3 months
7. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy
8. Self-reported or documented seropositivity for human immunodeficiency virus (HIV), hepatitis B natural infection (HBcAb positive serology), or hepatitis C
9. Known systemic hypersensitivity to any of the vaccine components (e.g. gold), or history of a life-threatening reaction to vaccines or to a vaccine containing any of the same substances
10. Current alcohol abuse or drug addiction (reported or suspected)
11. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
12. Thrombocytopenia or any coagulation disorder
13. Identified as an Investigator or employee of the Investigator or study centre with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (i.e. in the employment of the clinical trial sites).
14. Refusal to be informed if relevant results concerning the participant's health are revealed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety, tolerability and reactogenicity of the vaccine | 6 months following first vaccination or End Of Study (EOS), whichever is later
  Occurrence of solicited local reactogenicity signs and symptoms up to 7 days after each injection. Occurrence of solicited systemic reactogenicity signs and symptoms up to 14 days after each injection. Occurrence of unsolicited adverse events, serious adverse events (SAEs), and adverse events of special interest (AESI) up to 6 months following first vaccination or End Of Study (EOS), whichever is later.

SECONDARY OUTCOMES:
Assess the cellular immunogenicity of the vaccine candidate | 180 days following first vaccination
  Proportion of participants with T cells specific to PepGNP-COVID19 vaccine, and Proportion of subjects with activated cellular immunity cells via assessment of peptide-specific T cell response performed by cytometry, using dextramer staining and, by measuring activation markers upon stimulation with peptides
Assess the humoral immunogenicity of the vaccine candidate | 180 days following first vaccination
  For individuals seronegative at enrolment - Proportion of participants becoming seropositive (antibodies against SARS-CoV-2 as determined by Enzyme-linked Immunosorbent Assay (ELISA)), and For individuals seropositive at enrolment - Fold change in anti-SARS-CoV-2 antibodies as determined by Enzyme-linked Immunosorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto R Edison, MD, Principal Investigator — Research Institute for Tropical Medicine
Locations (2):
- Philippines (2):
  - Health Index Multispecialty Clinic, Barangay Toclong 2B, Imus, Cavite
  - Tropical Disease Foundation, Makati City, National Capital Region

IPD SHARING:
Plan to Share IPD: No